CLINICAL TRIAL: NCT00936949
Title: Posterolateral Surgical Approach Compared With Modified Lateral Approach: A Prospective, Randomised Trial
Brief Title: Posterolateral Surgical Approach Compared With Modified Lateral Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Kyung-Hoi, Koo professor, Seoul national University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNU 03-01
Record Dates: First submitted 2009-07-07; First posted 2009-07-10 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2009-07

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: total hip arthroplasty; posterolateral; modified lateral

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- posterolateral approach (Active Comparator): The posterolateral approach was described by many authors, but all share a common muscular interval in reference to the gluteus medius tendon. Using a gluteus maximus split, the posterolateral approach remains posterior to the gluteus medius and minimus. Exposure of the hip and proximal femur requires division of the posterior hip capsule and the external rotators. The exposure and dislocation are completed with flexion and internal rotation of the femur. After arthroplasty, the external rotators and posterior capsule was routinely repaired using a heavy absorbable suture.
  Interventions: Procedure: surgical approach
- modified lateral approach (Active Comparator): The operative technique described modified lateral approach as described by Mulliken et al.
  Interventions: Procedure: modified lateral approach

INTERVENTIONS:
Procedure: surgical approach — Using a gluteus maximus split, the posterolateral approach remains posterior to the gluteus medius and minimus. Exposure of the hip and proximal femur requires division of the posterior hip capsule and the external rotators. The exposure and dislocation are completed with flexion and internal rotation of the femur. After arthroplasty, the external rotators and posterior capsule was routinely repaired using a heavy absorbable suture.
  Other Names: posterolateral approach
  Arms: posterolateral approach
Procedure: modified lateral approach — The operative technique described modified lateral approach as described by Mulliken et al.
  Arms: modified lateral approach

SUMMARY:
It has been reported that the operative approaches have an effect on clinical outcome in total hip arthroplasty. The purpose of this prospective study was to compare clinical and radiological outcomes between anterolateral approach and posterolateral approach in total hip arthroplasty.

DETAILED DESCRIPTION:
Total hip arthroplasty is one of the most successful orthopaedic procedures for relieving pain and improving quality of life. But dislocation remains the leading early complication after total hip arthroplasty with a reported frequency between 0.4% and 11%. There are several risk factors of dislocation after total hip arthroplasty including patients, implants and surgical approaches. Among lots of risk factors, surgical approach has been debated as one of the important key factor influencing dislocation and abductor function. Direct lateral or posterolateral surgical approach is most commonly used in the total hip arthroplasty. The modified lateral approaches generally are thought to have lower dislocation rates and allow excellent acetabular exposure although limping is increased. The posterolateral approach may allow maintenance of abductor strength but it generally results in a higher dislocation rate. However, there are several reports that the posterolateral approach with capsular repair might be reduced dislocation rate.

We hypothesize the dislocation rate for the posterolateral approach with capsular repair is similar to modified lateral approaches for total hip arthroplasty. A prospective, randomized-controlled study was to examine the null hypothesis that the dislocation rate for the posterior approach with capsular repair was similar to modified lateral approaches for total hip arthroplasty at up to 2 year followup. We attempted to determine whether there was a difference in surgical parameters, component positioning, and clinical results of the modified lateral approach compared with the posterolateral approach.

ELIGIBILITY:
Inclusion Criteria:

* osteonecrosis
* primary or secondary osteoarthritis of the hips
* femoral neck fracture.

Exclusion Criteria:

* Patients with previous hemi- or total hip arthroplasty
* highly dislocated or severe ankylosed hip
* patients who are considered potentially unreliable or who may not reliably attend study visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2003-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
to examine the null hypothesis that the dislocation rate for the posterior approach with capsular repair was similar to modified lateral approaches for total hip arthroplasty at up to 2 year followup | up to 2 years

SECONDARY OUTCOMES:
to determine whether there was a difference in surgical parameters, component positioning, and clinical results of the modified lateral approach compared with the posterolateral approach. | Routine follow-up visits were scheduled for six weeks, three, six, nine, twelve months, and yearly thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Hoi Koo, professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul national University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea